CLINICAL TRIAL: NCT05387018
Title: The Effects of Hyperbaric Oxygen on Non-acute Traumatic Brain Injury
Status: Completed | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-0031
Record Dates: First submitted 2022-03-28; First posted 2022-05-24 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2023-03

CONDITIONS: Traumatic Brain Injury
Keywords: traumatic brain injury; hyperbaric oxygen; non-acute
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Observation group (hyperbaric oxygen + routine rehabilitation treatment): no special intervention
- control group (routine rehabilitation treatment): no special intervention

SUMMARY:
Traumatic brain injury (TBI) continues to be a major cause of death and disability throughout the world. The reduced cerebral blood flow secondary to the direct trauma-induced damage deregulates cerebral metabolism and depletes energy stores within the brain. Diffusion barriers to the cellular delivery of oxygen develop and persist. Besides, TBI often leads to intracranial hypertension, which in turn exacerbates diffusion disorders, further reducing cerebral oxygenation, and deteriorates the injury. By increasing the partial pressure of oxygen in blood, reducing intracranial pressure and cerebral edema, Hyperbaric oxygen therapy (HBO2) has been used in early treatment of TBI. However, due to the different severity of TBI, the clinical situation of early insult is complex and unpredictable, ordinarily there was a time delay between TBI and onset of HBO2 treatment averaging more than 2 weeks, especially in patients with severe TBI. Whether the delayed intervention is still effective is controversial.

DETAILED DESCRIPTION:
Traumatic brain injury (TBI) continues to be a major cause of death and disability throughout the world. The pathophysiological processes which occur post-TBI are complex and have not been fully elucidated. Penetrating injury, mechanical stress, cceleration-deceleration injury, and shear forces provide the direct trauma-induced damage. Subsequently, the reduced cerebral blood flow deregulates cerebral metabolism and depletes energy stores within the brain. Diffusion barriers to the cellular delivery of oxygen develop and persist. Besides, TBI often leads to intracranial hypertension, which in turn exacerbates diffusion disorders, further reducing cerebral oxygenation, and deteriorates the injury. Ischemia has been implicated as a major cause of secondary brain injury and death following severe brain injury.

Hyperbaric oxygen therapy (HBO2) has been used in early treatment of TBI. Studies have shown that increased tissue oxygen delivery is capable of driving an increase in oxygen utilization, leading to improved cerebral aerobic metabolism. By increasing the partial pressure of oxygen in blood, HBO2 increases cerebral oxygen saturation. In addition, HBO2 has been shown in both experimental and clinical studies to reduce intracranial pressure and cerebral edema after severe TBI. HBO2 has been shown to decrease mortality rates and improve functional outcome in severely brain-injured patients.

However, due to the different severity of TBI, the clinical situation of early insult is complex and diverse, and a considerable number of patients in the acute stage was accompanied by unstable intracranial hemorrhage, hemodynamic instability, ventilator assisted ventilation and other unpredictable conditions, therefore, ordinarily there was a time delay between TBI and onset of HBO2 treatment averaging more than 2 weeks, especially in patients with severe TBI. Whether the delayed intervention is still effective is controversial.

ELIGIBILITY:
Inclusion Criteria:

* The age ranges from 18 to 90
* Traumatic brain injury, Head CT scan confirmed the presence of at least one of the following findings: Intracranial hemorrhage, subdural hematoma, epidural hematoma, brain contusion, hemorrhagic brain contusion, subarachnoid hemorrhage, brain stem injury
* Those who had good compliance, signed informed consent and were eligible for inclusion according to the investigator's judgment.

Exclusion Criteria:

* Penetrating head injury
* Combined with spinal cord injury or peripheral nerve injury
* Severe coagulopathy
* Severe heart function, liver function, kidney function and other organ function abnormality
* The investigator considers the subject to be at potential risk or to have any other factors that may interfere with the subject

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who had been hospitalized for rehabilitation in our rehabilitation unit after traumatic brain injury, to study the differences in outcomes between those who received hyperbaric oxygen therapy within 3 months of injury and those who did not
Sampling Method: Non-Probability Sample
Enrollment: 390 (Actual)
Dates: Start 2022-03-31 (Actual); Primary Completion 2025-02-05 (Actual); Study Completion 2025-02-05 (Actual)

PRIMARY OUTCOMES:
Disability Rating Scale, DRS | 2014-2024
  Different points of DRS represent the degree of disability: 0 point : No; 1 point: Mild; 2-3 points: Partial; 4-6 points: Obvious; 7-11 points: Moderately severe; 12 to 16 points: Severe; 17-21 points: Extremely severe; 22-24: Vegetative state; 25-29 points: Extreme vegetative state; 30: Death
Glasgow Outcome Scale-Extend | 2014-2024
  The GOSE measures overall disability (independence, work, social and leisure activities, family and friendship and return to normal life) after TBI and divides patients into the following outcome categories:
  1= dead; 2 = vegetative state (VS); 3 = lower severe disability and complete dependence on others (Lower SD); 4 = upper severe disability and some dependency on others, but can be alone (on their own ) for 8 hours (Upper SD); 5= lower moderate disability, living independently, (not working or) working at a lower level of performance/sheltered work (Lower MD); 6 = upper moderate disability and returning to previous work with adjustments (Upper MD); 7 = lower good recovery with (almost back at full functional recovery) only minor physical or mental deficits (minor disability) (Lower GR);8 = upper good recoverythat implies full functional recovery (without any disability) (Upper GR)

SECONDARY OUTCOMES:
Glasgow Outcome Scale, GOS | 2014-2024
  The Glasgow Outcome Scale was divided into five scales, with poor prognosis at scales 1 to 3 and good prognosis at scales 4 to 5
Functional Independence Measure （FIM） | 2014-2024
  The FIM is composed of 18 items designed to operationally measure functional independence in self-care (eg, toileting), mobility (eg, walking, transfers), and cognition (eg, memory, communication, problem solving). Higher scores represent a greater level of independence.

CONTACTS AND LOCATIONS:
Overall Officials: Bing Xiong, master, Principal Investigator — director of department
Locations (1):
- The Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang Z, Li Z, Li S, Xiong B, Zhou Y, Shi C. Hyperbaric oxygen for moderate-to-severe traumatic brain injury: outcomes 5-8 years after injury. Med Gas Res. 2025 Mar 1;15(1):156-163. doi: 10.4103/mgr.MEDGASRES-D-24-00018. Epub 2024 Sep 25. PMID 39324933